CLINICAL TRIAL: NCT01400659
Title: The PIZZA-Salami Trial: Monocentric Randomised Cross-over Study of Carb Counting vs. Carb Plus Fat/Protein Counting Based Insulin Bolus Used for Sensor-augmented Continuous Subcutaneous Insulin Infusion (CSII) in Pediatric Patients
Brief Title: Pizza-Salami Study in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PPS2008
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: CSII; prandial insulin requirements; bolus calculation; dual-wave bolus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CARB Counting (Active Comparator): For CARB counting, insulin dose will be calculated according to the carbohydrate content of the test meal (1 carb unit = 10 g carbohydrate). The insulin-to-carbohydrate ratio will be applied according to the current individual therapy of the patient.
  Interventions: Procedure: CFP counting
- CFP counting (Active Comparator): For CFP counting, insulin dose will be calculated according the carbohydrate content (1 carb unit = 10 g carbohydrate) as well as fat/protein content (1 FPU = 100 kcal from fat and protein) of the meal. The insulin-to-carbohydrate ratio will be applied according to the current individual therapy of the patient. The insulin-to-FPU ratio is the same as the insulin to carb ratio.
  Interventions: Procedure: CARB counting

INTERVENTIONS:
Procedure: CFP counting — Patients receive a standardized test meal at lunch time. The required insulin dose is calculated by CFP counting. Insulin is given as bolus and basal rate using an insulin pump. Continuous glucose monitoring is performed by sensor-augmented pump system for 6 hours after the meal. The intervention is taking part under in-patient clinical conditions.
  Other Names: CFP algorithm according to Pankowska et al.
  Arms: CARB Counting
Procedure: CARB counting — Patients receive a standardized test meal at lunch time. The required insulin dose is calculated by CARB counting. Insulin is given as bolus and basal rate using an insulin pump. Continuous glucose monitoring is performed by sensor-augmented pump system for 6 hours after the meal. The intervention is taking part under in-patient clinical conditions.
  Other Names: CARB algorithm
  Arms: CFP counting

SUMMARY:
The Pizza-Salami-Study aims to investigate the efficacy of carbohydrate plus fat/protein (CFP) counting compared with carbohydrate (CARB) counting using normal and dual-wave bolus in sensor-augmented pump therapy in children and adolescents with type 1 diabetes. For fat/protein counting the model used by Pankowska et al. will be applied.

DETAILED DESCRIPTION:
This is a prospective, international multi-centre, open randomized clinical trial to assess whether the use of Paradigm REAL-Time System from the onset of Type 1 Diabetes (T1D) leads to a better glycaemic control after 12 months of T1D compared with the use of Paradigm 515/715 insulin pump combined with conventional Self-Monitoring Blood Glucose finger-sticks in paediatric patients. Total randomized treatment duration of the study for a patient will be 12 months with an optional phase of follow-up of 3 months.Patients eligible according to inclusion and exclusion criteria will be randomized to one of the two treatment groups. A total of 160 patients will be recruited. Each subject will participate in the study for 15 months, which includes 12 months of treatment and 3 months of follow-up. Each patient is asked to use either the Paradigm REAL-Time System that provides a combination of insulin pump and the Real-Time continuous glucose monitoring or Paradigm 515/715 insulin pump combined to conventional SMBG finger-sticks. Main time-points of assessments are at baseline (within one month after T1D onset) and 12 months thereafter. In total, there will be 6 study visits at the local site. During study, patients will regularly attend the outpatient clinic according to local Standard care, i.e. every 8±2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes
* Age 6 - 21 years
* Diabetes duration > 1 year
* Treatment with pump therapy (CSII) > 3 months
* Written informed consent by patients and parents
* Patients must be willing to wear a glucose sensor for two days and to perform capillary blood glucose measurement twice a day
* Patients must be willing to performed all study procedures

Exclusion Criteria:

* Language barriers
* Eating disorders
* Pregnancy
* Drug abuse
* Patient refutes participation or study procedures

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
CGM-Glucose Area Under the Curve | 6 hours after the test meal
  CGM = Continuous Glucose Monitoring

SECONDARY OUTCOMES:
Time of glucose nadir | 6 hours after the test meal
hyperglycemia (6h-AUC >180 mg/dl) | 6 h after the test meal
  AUC = Area Under the Curve
frequency and amount of interventional hypoglycemic therapy | 6 h after the test meal
  i.e. g of glucose required to treat hypoglycemia
frequency of adverse events (incl. SAE) | during hospitalization period of the study
  Hospital stay was from 2h before until 6h after teast meal. SAE = Severe Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Olga Kordonouri, MD, Principal Investigator — Kinderkrankenhaus auf der Bult

REFERENCES:
- [Background] Pankowska E, Blazik M. Bolus calculator with nutrition database software, a new concept of prandial insulin programming for pump users. J Diabetes Sci Technol. 2010 May 1;4(3):571-6. doi: 10.1177/193229681000400310. PMID 20513322
- [Derived] Kordonouri O, Hartmann R, Remus K, Blasig S, Sadeghian E, Danne T. Benefit of supplementary fat plus protein counting as compared with conventional carbohydrate counting for insulin bolus calculation in children with pump therapy. Pediatr Diabetes. 2012 Nov;13(7):540-4. doi: 10.1111/j.1399-5448.2012.00880.x. Epub 2012 Jul 6. PMID 22765260